CLINICAL TRIAL: NCT06984224
Title: Efficacy of Pulsed Direct Current Electrical Stimulation (Neubie) on Low Back Pain
Brief Title: Pulsed Direct Current Electrical Stimulation for Treatment of Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuFit - Neurological Fitness and Education (Industry)
Collaborators: EA Therapeutic Health (Unknown); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00086182
Record Dates: First submitted 2025-05-06; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Back Pain, Low
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Physical Therapy with adjunctive Neubie Pulsed Direct Current Device at 500 pps
  Interventions: Device: Neubie Direct Current Stimulation Device
- Control (No Intervention): Standard of Care Physical Therapy

INTERVENTIONS:
Device: Neubie Direct Current Stimulation Device — Pulsed Direct Current Electrical Stimulation Device
  Arms: Experimental

SUMMARY:
The goal of this interventional clinical trail is to determine the efficacy of the use of the Neubie pulsed direct current electrical stimulation device for the treatment of participants experiencing mechanical low back pain. The main question it aims to answer is:

Does treatment with the Neubie improve symptoms and time to resolution of back pain compared to standard of care?

Researchers will compare a 12 session treatment physical therapy regimen using the Neubie to standard of care to see if there is a difference in symptom severity and time to resolution.

Participants will:

* Visit the clinic 2 times a week to undergo active physical therapy treatments with or without electrical stimulation from the Neubie.
* Undergo testing and fill out surveys on evaluation and final session on quality of life, disability, pain, and spinal mobility.

DETAILED DESCRIPTION:
To determine the efficacy of direct current (DC) electrical stimulation (the Neubie device) on back pain, patients presenting with mechanical, non-radicular low back pain will enroll in a 4 to 6 week treatment regimen at EA Therapeutic Health. The first session will consist of an intake evaluation session that will include: Modified Oswestry Pain Scale, The Schober test for mobility, Heart Rate Variability, and Quality of Life Index. These tests will serve as baseline (and a within subject control) for the intervention.

Participants will then undergo a treatment protocol that incorporates either traditional physical therapy (PT) exercises (standard of care control) or PT exercises with the Neubie utilized concurrently (experimental group). Subjects will undergo an evaluation session prior to starting treatment that includes the Modified Oswestry Pain Scale, The Schober test for mobility, Heart Rate Variability, and Quality of Life Index.

The experimental group subjects will undergo 12 sessions of physical therapy over a 4 to 6-week period which include 45 min of various physical therapy exercises concurrently with the Neubie followed by a 15 minute passive Vagus nerve stimulation protocol with the Neubie.

Control group subjects will participate in a physical therapy protocol that includes manual therapy (e.g. trigger point release, mobilization of the sacroiliac (SI) joint and exercises for back strengthening and stretching. Experimental group subjects will participate in a physical therapy protocol that includes manual therapy (e.g. trigger point release, mobilization of the SI joint) and exercises for back strengthening and stretching in conjunction with Neubie DC e-stim. Both control and experimental groups will receive a customized Home Exercise Program with exercises to be performed at home 1 time a day.

ELIGIBILITY:
Inclusion Criteria:

1. Must show evidence of axial mechanical low back pain at least 3/10 on visual analog scale, without radiation to the lower limbs. Pain has to have been present for at least two weeks or diagnosed as chronic .
2. Normal lower limb strength
3. Able to attend twice weekly physical therapy visis for up to 6 weeks
4. 18 years of age, or older

Exclusion Criteria:

1. Currently pregnant
2. Cardiac pacemaker
3. Active or recently treated cancer
4. Active or recent blood clots
5. Epilepsy
6. Open wounds
7. History of lumbar spine fusion surgery
8. Radicular symptoms suggesting radiculopathy or spinal stenosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Modified Oswestry Disability Index | Pre-intervention
  MODIFIED OSWESTRY DISABILITY SCALE - Each question is scored from 0-5 (minimum to maximum). The point total from each section is summed and the then divided by the total number of questions answered and multiplied by 100 to create a percentage disability. The scores range from 0-100% with lower scores meaning less disability.
Modified Oswestry Disability Index | 6 weeks
  MODIFIED OSWESTRY DISABILITY SCALE - Each question is scored from 0-5 (minimum to maximum). The point total from each section is summed and the then divided by the total number of questions answered and multiplied by 100 to create a percentage disability. The scores range from 0-100% with lower scores meaning less disability.
Visual Analog Pain Scale | Pre-intervention
  The Visual Analog Scale (VAS) for measuring pain ranges from 0-10, with 0 representing "no pain" and 10 representing "worst pain imaginable".
Visual Analog Pain Scale | 6 weeks
  The Visual Analog Scale (VAS) for measuring pain ranges from 0-10, with 0 representing "no pain" and 10 representing "worst pain imaginable".
Schober Test | Pre-intervention
  Schober Test for Spinal Mobility
Schober Test | 6 weeks
  Schober Test for Spinal Mobility
Quality of Life Index | Pre-intervention
  Quality of Life Index Score has a range from 0 to 100. Lower values represent poorer quality of life, while higher values indicate better quality of life.
Quality of Life Index | 6 weeks
  Quality of Life Index Score has a range from 0 to 100. Lower values represent poorer quality of life, while higher values indicate better quality of life.
Heart Math HRV | Pre-intervention
  The Heart Math HRV system takes a reading of the participant's HRV. This is provided in a numerical value which will be used as the HRV "score".
Heart Math HRV | 6 weeks
  The Heart Math HRV system takes a reading of the participant's HRV. This is provided in a numerical value which will be used as the HRV "score".

CONTACTS AND LOCATIONS:
Overall Officials: Ramona von Leden, PhD, Study Director — NeuFit - Neurological Fitness and Education

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT06984224/Prot_SAP_000.pdf